CLINICAL TRIAL: NCT00268658
Title: Clinical Use of Andante SmartStep System in Gait Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: sor412805ctil
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2005-11

CONDITIONS: Ankle Injuries; Femoral Neck Fractures
Keywords: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Arthroscopy
MeSH Terms: conditions — Ankle Injuries; Femoral Neck Fractures

INTERVENTIONS:
Device: SmartStep(tm) biofeedback device

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the biofeedback gait training device in improving load bearing over an operated limb, during post-operative gait training therapy. The effectiveness of the device will also be tested in self-training at home.

DETAILED DESCRIPTION:
To evaluate the effectiveness of the biofeedback gait training device as a biofeedback training therapeutic tool in improving body-weight bearing over the affected lower limb, quality of gait, level of ambulation and physical independence during rehabilitation, in patients after orthopedic procedures during gait therapy training, and as a biofeedback device for self-training at home.

ELIGIBILITY:
Inclusion Criteria:

* Rehabilitation after operation
* Patient is allowed full weight bearing
* Patient is motivated and able to communicate and understands orders
* Patient is able to walk 10 meters
* Patient filled out agreement and consent form

Exclusion Criteria:

* Activity limitation due to medical disorder, medications, or emotional status.
* Pain markedly obstructs gait ability
* Documented peripheral neuropathy
* Functional limitation prior to the current condition
* Premorbid, ongoing major depression or psychosis
* Multiple/pathological fractures
* Serious early complications
* Terminally ill patients
* Pregnant women
* Participation in current or recent (within 60 days prior to surgery) clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
load bearing over the affected lower limb
quality/symmetry of gait
level of ambulation and physical independence

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Plotkin, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel